CLINICAL TRIAL: NCT06039943
Title: A Comparative Single Centre Study Assessing the Relationship Between Acoustic Breath Sounds as Measured by a Commercially Available Sound Recording Device Against Standard of Care (Spirometry) in the Assessment of Airflow Obstruction in Patients Who Plan to Undergo Spirometry Testing
Brief Title: Relationship Between Acoustic Breath Sounds and Spirometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Respiri US (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RKK7649
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Asthma COPD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Participants will undergo wheeze monitoring during tidal breathing prior to spirometry and during a spirometry test.
  Interventions: Device: Wheeze measurement

INTERVENTIONS:
Device: Wheeze measurement — Acoustic breath sounds will be measured during tidal breathing prior to spirometry and during a spirometry attempt.

SUMMARY:
The goal of this clinical trial is to assess whether wheeze as assessed by a commercially available wheeze monitor is comparable to lung function as measured during a spirometry test. The main questions it aims to answer are whether measures of airflow obstruction (FEV1, FEV1/FVC, PEF) correlate with wheeze score (Tw/Ttot%).

Participants consenting to take part will undergo wheeze measurement prior to and during a spirometry test and will be asked to complete a series of symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adult (aged 18-95) University Hospitals Birmingham patient's attending the Lung Function and Sleep Department (LF&S) routinely as part of their standard clinical management pathway for Lung Function testing that includes Spirometry assessments.
* All patients irrespective of condition will be approached to participate.

Exclusion Criteria:

* Subjects who are contraindicated to perform spirometry on the day of testing
* Subjects who cannot speak or read English
* Patients accessing non-adult services
* Subjects who are unable or do not wish to consent
* Patients with known or suspected restrictive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Wheeze score (Tw/Ttot%) | Day 1
  The average proportion of each breath that contained wheeze during a 30 second breath sound recording.
FEV1/FVC | Day 1
  the ratio between forced expiratory volume in the first second (FEV1) and forced vital capacity (FVC)
FEV1 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Richard Glover, Principal Investigator — University Hospitals Birmingham
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers